CLINICAL TRIAL: NCT03796702
Title: Early Versus Late Closure of Preventive Ileostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High postoperative morbidity rate
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Rimantas Bausys, Investigator, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-12-30; First posted 2019-01-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ileostomy, Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early closure of preventive ileostomy (Experimental): A preventive ileostomy is closed 30 days after the primary surgery
  Interventions: Procedure: Deileostomy
- Late closure of preventive ileostomy (Experimental): A preventive ileostomy is closed 90 days after the primary surgery
  Interventions: Procedure: Deileostomy

INTERVENTIONS:
Procedure: Deileostomy — Deileostomy

SUMMARY:
The study is designed and performed as a prospective randomized controlled single-center study. Patients who underwent rectal resection with preventive ileostomy due to rectal cancer will be included. The study investigates the effect of reversing a temporary ileostomy after 30 vs 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with temporary ileostomy after rectal resection for rectal cancer
* Patients willing to participate in the study

Exclusion Criteria:

* Anastomosis insufficiency detected clinically or radiologically.
* Patients, who are physically and mentally unfit to undergo surgery or to be followed-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | 30 days after surgery
  Patients are scored according to the Clavien-Dindo Classification of Surgical Complications.

SECONDARY OUTCOMES:
Hospitalization time after ileostomy closure | 30 days after surgery
  Hospitalization time
30-days re-admission rate | 30 days after surgery
  Re-admission rate during 30 days after re-admission
Quality of life of patients after ileostomy closure | at 3, 6, 9 and 12 moths after surgery
  Patients quality of life is assessed with EORTC QLQ-C30 questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided